CLINICAL TRIAL: NCT04571671
Title: Do müllerian Anomalies Affect Embryo Implantation?
Acronym: AM
Status: Completed | Type: Observational
Sponsor: IVI Vigo (Other)
Collaborators: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Other Study IDs: 1405-VIG-029-EM
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Uterine Diseases
MeSH Terms: conditions — Uterine Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Women with Müllerian anomalies who have received an oocyte donation. The diagnosis of Müllerian anomalies is established when a cavity is demonstrated uterine abnormality with any of the defects described in the American classifications or European in transvaginal ultrasound, hysteroscopy or hysterosalpingography (HSG). The differential diagnosis in case of doubts is established with 3D ultrasound, MRI or hystero / laparoscopy. All the septa have been resected prior to performing the OVODON cycle.
  Interventions: Other: Collect retrospectively data
- Control group: Patients who receive donated oocytes and who do not present Müllerian anomalies. An absence of AM, a transvaginal ultrasound, an HSG or a normal hysteroscopy with a uterine cavity with a normal shape and absence of intracavitary images is considered
  Interventions: Other: Collect retrospectively data

INTERVENTIONS:
Other: Collect retrospectively data — Analyse the incidence of Mullerian anomalies in these populations

SUMMARY:
Müllerian anomalies (MA) are associated with infertility and affect approximately 6.3% of the infertile population. The estimation of the frequency of MAs is not without controversy because it depends on the diagnostic method used and sometimes on the established diagnostic criteria. This pathology is associated with abortion during the second trimester in addition to other complications that include preterm labor, fetal malpositions and an increased rate of caesarean section, although some patients may remain asymptomatic. An association between MA and endometriosis has been described and in particular the case of the septum uterus, therefore it is difficult to establish whether the reproductive results of women with MA tdepend only on the uterine factor or also on the quality of the oocytes.

DETAILED DESCRIPTION:
The main reproductive problems associated with these malformations include, abortion , recurrent abortion ectopic pregnancy and preterm delivery . The experience gained from oocyte donation shows that these women are pregnant less, even with the transfer of good quality embryos. The hypothesis of this poor uterine receptivity is in the poor endometrial vascularization that can decrease embryo implantation. The reason for infertility in women with AM includes decreased muscle mass, decreased endometrial vascularization, decreased capacity of the endometrial cavity, less receptive areas (septum). The lower fertility observed in some women with Müllerian malformations has been partially explained by its tubal factor and its association with endometriosis, with a higher prevalence in them, compared to patients without malformations.

Studies have confirmed an irregular differentiation and estrogenic maturation of the endometrium lining the uterine septum or its internal structure, which has less presence of connective tissue and more muscle mass. Given the confusion generated if the unfavorable reproductive result is due to oocyte quality or endometrial receptivity, it is necessary to use a model that guarantees oocyte / embryo quality and this is offered by oocyte donation. The aim is to evaluate the implantation rate in women with MA who receive donated oocytes compared to women without MA.

ELIGIBILITY:
Inclusion Criteria:

* Women included in the oocyte donation program at IVI Vigo and Valencia 2000-2019.
* Sperm count greater than 1,000,000 per ml.
* Transfer on day 5 of embryo development of at least one good quality embryo.

Exclusion Criteria:

* Testicular biopsy.
* Any indication for preimplantation genetic diagnosis or screening.
* Uterine fibroid greater than 4 cm.
* Presence of ultrasound or diagnosis by HSG or laparoscopy of hydrosalpinx uni or bilateral.
* Recurrent abortion.
* Any abnormality of the uterine cavity other than MA: submucosal myoma, endometrial polyp, or uterine synechiae.

Ages: 35 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Women with Müllerian anomalies who have received an oocyte donation. The diagnosis of Müllerian anomalies is established when a cavity is demonstrated uterine abnormality with any of the defects described in the American classifications or European in transvaginal ultrasound, hysteroscopy or hysterosalpingography (HSG). The differential diagnosis in case of doubts is established with 3D ultrasound, MRI or hystero / laparoscopy. All the septa have been resected prior to performing the OVODON cycle.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2014-01-20 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-07-25 (Actual)

PRIMARY OUTCOMES:
embryo implantation rate | Since 2000 to april 2019
  To compare embryo implantation rate

CONTACTS AND LOCATIONS:
Overall Officials: Ekin DR Muñoz, MD, Principal Investigator — IVI Vigo; Agustina Ramos Gutierrez, Study Chair — IVI Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makino T, Umeuchi M, Nakada K, Nozawa S, Iizuka R. Incidence of congenital uterine anomalies in repeated reproductive wastage and prognosis for pregnancy after metroplasty. Int J Fertil. 1992 May-Jun;37(3):167-70. PMID 1355763
- [Derived] Munoz E, Fernandez I, Pellicer N, Mariani G, Pellicer A, Garrido N. Reproductive outcomes of oocyte donation in patients with uterine Mullerian anomalies. Fertil Steril. 2023 Oct;120(4):850-859. doi: 10.1016/j.fertnstert.2023.06.029. Epub 2023 Jun 29. PMID 37392783